CLINICAL TRIAL: NCT03160768
Title: Feasibility of Isolating P16 Expression
Status: Completed | Type: Observational
Sponsor: St. Jude Children's Research Hospital (Other)
Collaborators: Sapere Bio (Industry)
Responsible Party: Sponsor
Other Study IDs: HPP21
Record Dates: First submitted 2017-05-18; First posted 2017-05-19 (Actual); Last update posted 2019-05-06 (Actual); Status verified 2019-05

CONDITIONS: Childhood Cancer
Keywords: p16; T cell isolation; physiologic age
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood specimen.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Expression of the cell cycle regulator p16INK4a increases with age and toxic stressors. In mice, both radiation and chemotherapy are known to increase p16. Due to its influence on age-related regenerative capacity, p16 is an excellent candidate biomarker of physiologic reserve that may identify patients able to withstand the stressor of chemotherapy (low p16) from those unlikely to tolerate chemotherapy (high p16). That is, expression of p16 may predict physiologic, rather than chronologic, age. Such findings could have implications for care of cancer survivors and treatment decision-making in cancer patients.

STUDY OBJECTIVE: This is an observational pilot study to determine the feasibility of isolating p16INK4a in CD3+ T lymphocytes in adults treated with chemotherapy for cancer during childhood.

DETAILED DESCRIPTION:
At St. Jude Children's Research Hospital, survivors who meet the eligibility criteria will be identified from SJLIFE protocol participants. After signing consent, the subject will have a blood specimen collected at the same time as the blood draw for the SJLIFE protocol. These samples will have T cell isolation performed then placed on ice and stored until batch shipment for investigation of p16 expression.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled in the SJLIFE study at St. Jude children's Research Hospital.
* Survivor of childhood cancer.
* Is 18 years of age and older.
* No evidence of cancer recurrence.
* Received prior chemotherapy (prior radiotherapy is allowed).

Exclusion Criteria:

* Inability or refusal to give consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be childhood cancer survivors enrolled in the long-term follow-up study at St. Jude Children's Research Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 85 (Actual)
Dates: Start 2017-05-25 (Actual); Primary Completion 2019-05-02 (Actual); Study Completion 2019-05-02 (Actual)

PRIMARY OUTCOMES:
Number of samples with successful isolation of expression of p16INK4a in CD3+ T lymphocytes | Within 3 months of enrollment of the last participant
  Blood samples will be drawn once at a regularly scheduled follow-up visit. After T cells are isolated, the samples will be sent in one batch for further processing and investigation of p16 expression.

CONTACTS AND LOCATIONS:
Overall Officials: Kirsten K. Ness, PT, PhD, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St. Jude Children's Research Hospital — http://www.stjude.org/protocols